CLINICAL TRIAL: NCT03341585
Title: Influence of Expiration Lente Prolongée on Gastro-oesopageal Reflux in Infants Under the Age of 1 Year
Brief Title: Influence of Expiration Lente Prolongée on Gastro-oesophageal Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Filip Van Ginderdeuren, Prof.Dr., Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVG005
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Gastro-esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expiration Lente Prolongée (Experimental): In this controlled trial with intra-subject design infants will be studied using multichannel intraluminal impedance pH (pH-MII) monitoring , during which they receive one 20 min session of 'Expiration Lente Prolongée (ELPr)' . The number of reflux episodes (RE) is the outcome measure. The results obtained during and 20 min after the intervention will be compared to a period of 20 min before treatment ( control ).
  Interventions: Other: expiration lente prolongée

INTERVENTIONS:
Other: expiration lente prolongée — l'Expiration Lente Prolongée (ELPr) is a passive technique to enhance the expiration used in infants, obtained by a slow and increasing manual thoraco-abdominal pression applied at the end of a spontaneous expiration till the residual volume. The aim is to obtain a bigger expired volume compared to a normal expiration and drain the mucus out of the airways (Postiaux 2003). This technique has been invented by Guy Postiaux and is used in the Chest Physiotherapy (CPT).

SUMMARY:
The purpose of this study is to determine whether a specific airway clearance technique, l'Expiration Lente Prolongée (ELPr), induces or aggravates gastro-oesophageal reflux in infants under the age of one year. Infants referred to hospital for a multichannel intraluminal impedance pH (pH-MII) monitoring are included in this study. Participation is only possible after signing the informal consent by one of the parents.

ELIGIBILITY:
Inclusion Criteria:

* Infants under the age of one year and on suspicion of GOR who were referred for 24h impedance-pH monitoring are included in this study.

Exclusion Criteria:

* prematurity (gestational age less than 37 weeks),
* the use of anti-reflux medication and reflux surgery (Nissen fundoplication)

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
number of refluxes | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: filip van ginderdeuren, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lievens L, Vandenplas Y, Vanlaethem S, Van Ginderdeuren F. Prolonged Slow Expiration Technique and Gastroesophageal Reflux in Infants Under the Age of 1 Year. Front Pediatr. 2021 Sep 8;9:722452. doi: 10.3389/fped.2021.722452. eCollection 2021. PMID 34568241